CLINICAL TRIAL: NCT00404261
Title: An Open Label, Multicentre Study to Evaluate Patient Satisfaction With Fluticasone/Salmeterol HFA MDI With Counter in Adult Subjects (18 Years of Age and Older) With Asthma or COPD.
Brief Title: Evaluation Of Patient Satisfaction Of Metered Dose Inhaler (MDI) With Counter In Asthmatics And Chronic Obstructive Pulmonary Disease Patients (COPD).
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 108835
Record Dates: First submitted 2006-11-27; First posted 2006-11-28 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Asthma
Keywords: Fluticasone Propionate; healthcare professional satisfaction; patient satisfaction; metered dose inhaler with counter; Salmeterol; Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Asthma; Patient Satisfaction; Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Other): Fluticasone/Salmeterol HFA MDI without counter
  Interventions: Drug: Fluticasone/Salmeterol HFA
- Arm 2 (Other): Fluticasone/Salmeterol HFA MDI with counter
  Interventions: Drug: Fluticasone/Salmeterol HFA

INTERVENTIONS:
Drug: Fluticasone/Salmeterol HFA — Fluticasone/Salmeterol HFA, 2 puffs twice daily

SUMMARY:
The purpose of this study is to evaluate the level of satisfaction experienced by asthma or chronic obstructive pulmonary disease (COPD) patients when using the Fluticasone/Salmeterol HFA Metered Dose Inhaler (MDI) with counter, as compared to using Fluticasone/Salmeterol HFA MDI without counter.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient
* Documented physician diagnosis of asthma or COPD
* Requires use of a controller and long acting beta 2 agonist
* Ability to provided written informed consent

Exclusion Criteria:

* Patients with life threatening asthma or COPD
* Historical or current evidence of significant diseases
* Immediate or delayed hypersensitivity to inhaled short acting beta2agonist or sympathomimetic drug or any component of the MDI formulation
* History of drug or alcohol abuse Abnormal chest x ray not consistent with asthma or COPD
* Use of supplemental oxygen; systemic corticosteroids; short acting beta2agonists other than VENTOLIN HFA; antibiotics for respiratory infections; anti-arrhythmics; anticonvulsants; central nervous system stimulants; tricyclic antidepressants and monoamine oxidase inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2007-01; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction questionnaires administered at baseline and at the end of treatment (day 30). | Day 30

SECONDARY OUTCOMES:
Healthcare professional satisfaction questionnaires administered at baseline and at the end of treatment (day 30) Patient compliance as measured by the device counter readings at the end of treatment (day 30), compared to the baseline reading. | Day 30
Healthcare professional satisfaction questionnaires Patient Compliance Safety Evaluations: adverse events | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Australia (4):
  - GSK Investigational Site, Auchenflower, Queensland
  - GSK Investigational Site, Caboolture, Queensland
  - GSK Investigational Site, Kippa-Ring, Queensland
  - GSK Investigational Site, Perth, Western Australia